CLINICAL TRIAL: NCT02651077
Title: Looking for a Link Between Endometriosis and Exposure to Lipophilic Environmental Chemicals Like Brominated Flame Retardant (ENDOTOX Study)
Brief Title: Endometriosis and Brominated Flame Retardant (ENDOTOX Study)
Acronym: ENDOTOX
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: ONIRIS (Industry)
Responsible Party: Sponsor
Other Study IDs: RC13_0380
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Endometriosis
Keywords: Endometriosis, chemical contaminants, BFRs
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — omental adipose tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Group: 38 women with severe and deep endometriosis, aged 18 to 45 years old and hospitalized at Nantes University Hospital for surgical indication of endometriosis lesions ablation.
- Control Group: 38 women aged 18 to 45 years old without suggestive signs of endometriosis

SUMMARY:
The investigators wish to highlight, in a Case-Control design, if there is an increased concentration of BFRs in omental adipose tissue of cases ( women with severe endometriosis with surgical indication ) versus bioaccumulation recorded in a control cohort ( women recruited in obstetrics and gynecology or visceral surgery showing no sign of endometriosis ) . Pairing will be operate on Age (+/- 5 years compared to the case ) , BMI ( BMI 5 Classes described by the HAS) and previous breastfeeding experience (yes / no , opposite the release expected bioaccumulate contaminants in breast adipose tissue , when the lactation ) .

ELIGIBILITY:
Inclusion criterion for de cases :

* Age : 18-45 years old
* Deep endometriosis with or without endometriomas that need surgery (clinical examination, MRI, surgery)
* Accessing to the omental and/or parietal adipose tissue
* Non opposition of the patients for the samples collection and consent for the present study.

Inclusion criterion for the controls :

* Patients without any history of endometriosis and without suggestive symptomatology. Often patients operated for cesarean section.
* Possible access to the adipose tissue of the omentum or abdominal wall

Exclusion criterion for the cases :

* Pregnancy
* Death

Exclusion criterion for controls :

* Pregnancy
* Death

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 38 women with severe and deep endometriosis, aged 18 to 45 years old and hospitalized at Nantes University Hospital for surgical indication of endometriosis lesions ablation.
  And 38 women aged 18 to 45 years old without suggestive signs of endometriosis
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Concentrations of brominated flame retardant (BFR) in adipose tissue and serum | baseline

SECONDARY OUTCOMES:
Concentrations of dioxins in adipose tissue and serum | baseline
Concentrations of polychlorinated biphenyls (PCBs), | baseline
Concentrations of organochlorine pesticides (OCPs) in adipose tissue and serum | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephane PLOTEAU, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France